CLINICAL TRIAL: NCT05579509
Title: Personalizing Preprocedural Sedation for Regional Anesthesia: a Randomized Trial and Qualitative Assessment of Patient-Centered Outcomes and Experience
Brief Title: Personalizing Preprocedural Sedation for Regional Anesthesia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Yun-Yun K. Chen, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022P001901
Record Dates: First submitted 2022-09-29; First posted 2022-10-13 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Catastrophizing Pain
Keywords: Catastrophizing; Regional anesthesia; Nerve block; Preprocedural sedation
MeSH Terms: interventions — Midazolam; Fentanyl

STUDY DESIGN:
Intervention Model Description: Parallel and crossover design. Subjects in Arm 2 may crossover to Arm 1 if they receive pharmacologic sedation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High Pain Catastrophizing (Experimental): Based on the Pain Catastrophizing Scale (PCS)
  Interventions: Drug: Midazolam and Fentanyl; Behavioral: Educational Reassurance
- Low Pain Catastrophizing (Experimental): Based on the Pain Catastrophizing Scale (PCS)
  Interventions: Drug: Midazolam and Fentanyl; Behavioral: Educational Reassurance

INTERVENTIONS:
Drug: Midazolam and Fentanyl — Prior to the start of the nerve block, patients in Arm 1 will receive titrated pharmacological sedation with IV midazolam with a goal of achieving moderate sedation. If pain is felt despite subcutaneous lidocaine, IV fentanyl may be administered with a goal of achieving moderate sedation with analgesia.
  Other Names: Versed; Sublimaze
Behavioral: Educational Reassurance — Patients in the nonpharmacologic group will receive intraprocedural education and reassurance without pharmacologic sedation. They will have the option to receive more pharmacologic sedation at any point during the nerve block (cross-over to titrated sedation group).

SUMMARY:
This is a prospective, randomized study in patients who receive a nerve block prior to surgery. The aim is to investigate whether individual differences in psychosocial and pain profiles may play a role in how patients experience sedation for regional anesthesia. The study will utilize a mixed-methods approach, including a randomized controlled intervention and semi-structured interviews, in order to systematically investigate the relationship between an individual patient's level of catastrophizing and efficacy of procedural sedation, while exploring patient satisfaction with the preoperative nerve block experience.

DETAILED DESCRIPTION:
The primary quantitative outcome will be pain severity during nerve block placement. Secondary quantitative outcome is patient satisfaction. Validated psychometric assessment tools (pain catastrophizing scale) will be used to stratify patients according to baseline degree of pain catastrophizing (high versus low baseline pain catastrophizing). These groups will then be randomized to receive either titrated pharmacologic sedation (i.e., additional midazolam and fentanyl beyond a standard low midazolam dose) or intraprocedural educational reassurance. Semi-structured interviews and qualitative analysis will be used to explore patient's experiences with nerve block placement and identify themes regarding what makes this experience more positive or negative for individuals with different characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18
* English speaking
* Willingness to undergo psychophysical testing
* Willingness to have nerve block performed
* Surgical or procedural patient
* Single shot nerve block

Exclusion Criteria:

* Cognitive dysfunction that precludes communication
* Declines or is not eligible clinically to receive sedation with midazolam and/or fentanyl at discretion of the non-study clinical team (Examples: frailty, cognitive dysfunction)
* Allergy or hypersensitivity to midazolam or fentanyl
* Declines nerve block
* Does not complete survey needed for randomization
* Current pregnancy and/or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-10-22 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Pain scale | Immediately following procedure
  Procedural pain rating during the nerve block procedure on a 0 (no pain) to 10 (severe pain) Likert scale. Higher scores represent a worse outcome.

SECONDARY OUTCOMES:
Patient satisfaction | Immediately following procedure
  Satisfaction with nerve block on a 1 (low satisfaction) to 10 (high satisfaction) Likert scale. Higher scores represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Yun K Chen, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chen YK, Wilson JM, Gokul SR, Collins PW, Kiik M, Vlassakov K, Schreiber KL. Education or sedation? A randomized clinical trial of impact on procedural pain and satisfaction during regional block placement, and the moderating effect of pain catastrophizing. Reg Anesth Pain Med. 2025 Jun 5:rapm-2025-106644. doi: 10.1136/rapm-2025-106644. Online ahead of print. PMID 40473409